CLINICAL TRIAL: NCT03618095
Title: REPRISE IV: REpositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of LOTUS Edge Valve System in IntermediatE Surgical Risk Subjects
Brief Title: REPRISE IV: LOTUS Edge Valve System in Intermediate Surgical Risk Subjects
Acronym: REPRISE IV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational Medical Device is no longer available
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2354
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Evaluation of Lotus Edge to treat patients with aortic stenosis. A single intervention is being evaluated in 3 study arms, the roll-in, main and bicuspid cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Main Cohort (Experimental): Transcatheter Aortic Valve Replacement (TAVR) with the LOTUS Edge Valve System
  Interventions: Device: LOTUS Edge Valve System
- Roll-In Cohort (Experimental): Transcatheter Aortic Valve Replacement (TAVR) with the LOTUS Edge Valve System
  Interventions: Device: LOTUS Edge Valve System
- Bicuspid Cohort (Experimental): Transcatheter Aortic Valve Replacement (TAVR) with the LOTUS Edge Valve System
  Interventions: Device: LOTUS Edge Valve System

INTERVENTIONS:
Device: LOTUS Edge Valve System — TAVR with the LOTUS Edge Valve System

SUMMARY:
REPRISE IV: REpositionable Percutaneous Replacement of Stenotic Aortic Valve through Implantation of LOTUS Edge Valve System in IntermediatE Surgical Risk Subjects

DETAILED DESCRIPTION:
To evaluate safety and effectiveness of the LOTUS Edge™ Valve System when used with the Lotus™ or iSleeve™ Introducer Sets for transcatheter aortic valve replacement (TAVR) in symptomatic subjects with severe aortic stenosis who are considered at intermediate risk for surgical valve replacement including those who have a bicuspid native valve.

ELIGIBILITY:
Inclusion Criteria:

* Subject has documented severe aortic stenosis defined as initial aortic valve area (AVA) ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2) AND a mean pressure gradient ≥40 mm Hg OR maximal aortic valve velocity ≥4.0 m/s OR Doppler velocity index ≤0.25 as measured by echocardiography and/or invasive hemodynamics. Note: In cases of low flow, low gradient aortic stenosis with left ventricular dysfunction (ejection fraction <50%), dobutamine can be used to assess the grade of aortic stenosis (maximum dobutamine dose of 20 mcg/kg/min recommended)c; the subject may be enrolled if echocardiographic criteria are met with this augmentation. (IC1)
* A subject in the Bicuspid Aortic Valve Nested Registry cohort must have a documented Sievers Type 0 or Sievers Type 1 bicuspid aortic valve based on computed tomography (CT) assessment and confirmed by the CT core lab with hemodynamic parameters that meet the criteria in IC1.
* Subject has a documented aortic annulus size of ≥20 mm and ≤27 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]).
* Subject has symptomatic aortic valve stenosis per IC1 definition above with New York Heart Association (NYHA) Functional Class ≥ II.
* Heart team (which must include an experienced cardiac interventionalist and an experienced cardiac surgeon) agrees that the subject is at intermediate risk of operative mortality (≥3% and <8% at 30 days based on the Society of Thoracic Surgeons [STS] risk score and other clinical comorbidities unmeasured by the risk calculator) and TAVR is appropriate. Note: Risk of operative mortality must be assessed via an in-person evaluation by a center cardiac surgeon and must be confirmed by the CRC (which must include an experienced cardiac surgeon).
* Heart team agrees that the subject is likely to benefit from valve replacement. IC7. Subject (or legal representative) has been informed of the study requirements and the treatment procedures, and provides written informed consent.
* Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow-up visits.
* Subject is expected to be able to take the protocol-required adjunctive pharmacologic therapy.

Exclusion Criteria:

* Subject has a unicuspid or bicuspid aortic valve (not applicable to subjects in the Bicuspid Nested Registry cohort).
* Subjects in the Bicuspid Nested Registry cohort will have a documented Sievers Type 0 or Sievers Type 1 bicuspid aortic valve based on CT assessment and confirmed by the CT core lab. Subjects are not eligible for inclusion in the Bicuspid Nested Registry cohort if the maximum diameter of the ascending aorta is >45 mm or if the subject has another indication for aortic root replacement. Subjects with a Sievers Type 2 bicuspid valve are not eligible for enrollment in any study cohort.
* Subject has had an acute myocardial infarction (MI) within 30 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total creatine kinase (CK) elevation ≥ twice normal in the presence of creatine kinase-myoglobin band (CK-MB) elevation and/or troponin elevation).
* Subject has had a cerebrovascular accident or transient ischemic attack clinically confirmed by a neurologist or neuroimaging within the past 6 months prior to study enrollment.
* Subject is on renal replacement therapy or has Glomerular Filtration Rate (GFR) <20 (based on hospital preferred method). See AEC1 below if subject is in the CT Imaging Substudy.
* Subject has a pre-existing prosthetic aortic or mitral valve.
* Subject has severe (4+) aortic, tricuspid, or mitral regurgitation.
* Subject has moderate to severe mitral stenosis (mitral valve area ≤1.5 cm2 and diastolic pressure half-time ≥150 ms, Stage C or Dc).
* Subject has a need for emergency surgery for any reason.
* Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.
* Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.
* Subject has platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
* Subject will refuse transfusions or has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen.
* Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all P2Y12 inhibitors, heparin, nickel, tantalum, titanium, or polyurethanes.
* Subject has a life expectancy of less than 24 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment.
* Subject has hypertrophic cardiomyopathy.
* Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty or pacemaker or implantable cardioverter defibrillator implantation, which are allowed).
* Subject has multivessel coronary artery disease with a Syntax score >22, and/or an unprotected left main coronary artery.
* Subject has severe left ventricular dysfunction with ejection fraction <20%.
* Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
* Subject has arterial access that is not acceptable for the study device delivery system as defined in the device Instructions For Use.
* Subject has severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely; marked tortuosity; significant narrowing of the abdominal aorta; severe unfolding of the thoracic aorta; or thick, protruding, ulcerated atheroma in the aortic arch).
* Subject has current problems with substance abuse (e.g., alcohol, etc.) that may interfere with the subject's participation in this study.
* Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
* Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation. Enrollment is permissible after permanent pacemaker implantation.
* Subject has severe incapacitating dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher U. Meduri, MD, MPH, Principal Investigator — Piedmont Heart Institute; Vinod H. Thourani, MD, Principal Investigator — Piedmont Heart Institute
Locations (50):
- United States (49):
  - Huntsville Hospital, Huntsville, Alabama
  - Tucson Medical Center, Tucson, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Mills-Peninsula Medical Center - Sutter Health, Burlingame, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC Medical Center, Los Angeles, California
  - Saint Joseph Hospital, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Medstar Heart and Vascular Institute, Washington D.C., District of Columbia
  - JFK Medical Center, Atlantis, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Wellstar Research Institute, Marietta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana University Health - Methodist Hospital, Indianapolis, Indiana
  - Via Christi Hospital, Wichita, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Charlton Memorial Hospital - Southcoast Health, Fall River, Massachusetts
  - Spectrum Health - Grand Rapids, Grand Rapids, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Englewood Hospital, Englewood, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU Winthrop Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center/NewYork Presbyterian Hospital, New York, New York
  - Novant Health Heart & Vascular Institute - Charlotte, Charlotte, North Carolina
  - UNC Rex Hospital, Raleigh, North Carolina
  - The Lindner Center for Research and Education, Cincinnati, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Memorial Hospital - Prisma Health, Greenville, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Memorial Hermann - Texas Medical Center, Houston, Texas
  - University of Texas - Memorial Hermann Southwest, Houston, Texas
  - Baylor Scott & White The Heart Hospital, Plano, Texas
  - Inova Fairfax Hospital, Annandale, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - WVU Heart & Vascular Institute, Morgantown, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert Hospital - Medical College of Wisconsin, Milwaukee, Wisconsin
- Monash Cardiovascular Research Centre, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated early. Enrollment was stopped before the target number of subjects were enrolled to achieve target power and was insufficient to produce statistically reliable results. All characteristics are based on the total enrollment and not the individual arms as there were not sufficient subjects. In addition, as there was not sufficient power, and even the enrolled subjects did not all reach 1 year follow-up, no primary endpoint analysis was warranted.
Groups:
- Roll-In Cohort: Transcatheter Aortic Valve Replacement (TAVR) with the LOTUS Edge Valve System for sites that do not have implantation experience with the LOTUS Edge Valve System. At least 2 per site needed.
  LOTUS Edge Valve System: TAVR with the LOTUS Edge Valve System
- Bicuspid Cohort: Transcatheter Aortic Valve Replacement (TAVR) with the LOTUS Edge Valve System in a native bicuspid aortic valve.
  LOTUS Edge Valve System: TAVR with the LOTUS Edge Valve System
Period: Overall Study
Arm/Group | Main Cohort | Roll-In Cohort | Bicuspid Cohort
Started | 274 | 63 | 45
Completed | 0 | 0 | 0
Not Completed | 274 | 63 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Cohort | Roll-In Cohort | Bicuspid Cohort | Total
Number analyzed (Participants) | 274 | 63 | 45 | 382
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (6.1) | 79.8 (6.8) | 74.8 (6.1) | 77.7 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 30 | 22 | 179
  Male | 147 | 33 | 23 | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — More than one category can be selected per subject if desired.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 1
    Black, of African heritage | 14 | 3 | 1 | 18
    Caucasian | 250 | 54 | 43 | 347
    Hispanic or Latino | 5 | 3 | 1 | 9
    Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
    Other | 3 | 2 | 1 | 6
    Not Disclosed | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 257 | 63 | 42 | 362
  Australia | 17 | 0 | 3 | 20
Society of Thoracic Surgeons (STS) Risk Score [Mean (Standard Deviation); unit: Percent %] — Measure Description: The Society of Thoracic Surgeons Score is a risk model used to predict a subject's risk of mortality and morbidities for the most commonly performed cardiac surgeries. The model is a percentage score from 0 to 100 where a lower score means a lower risk and higher score means a higher risk.
  Percent % | 2.6 (1.1) | 3.4 (2.1) | 2.1 (0.9) | 2.7 (1.4)
European System for Cardiac Operative Risk Evaluation (EuroSCORE) [Mean (Standard Deviation); unit: Percent predicted] — Measure Description: The European System for Cardiac Operative Risk Evaluation is a risk model where if a risk factor is present in a subject, a weight or number is assigned. The weights are added to give an approximate percent predicted mortality. A higher score means a higher risk and a lower score means a lower risk.
  Percent predicted | 2.6 (1.9) | 3.0 (2.5) | 2.4 (2.1) | 2.6 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Composite of All-cause Mortality and All Stroke.
Description: Pre-specified primary outcome measure in the protocol for the Main Cohort only. Critical safety events that are observed in the elderly population undergoing TAVR; assessments recommended by Valve Academic Research Consortium (VARC)
Time Frame: 1 year post index procedure and device implantation
Population: This study was terminated early. Enrollment was stopped before the target number of subjects were enrolled. Additionally, patient follow-up was terminated therefore, not all enrolled subjects at the time of termination were followed through the Primary Endpoint timepoint (1 Year). This analysis only represents those patients who reached 1 year at the time of study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Cohort
Number analyzed (Participants) | 174
Participants | 18

ADVERSE EVENTS:
Time Frame: Events collected through the Termination of the study, majority of patient an average of 30 days.
Arm/Group | Main Cohort | Roll-In Cohort | Bicuspid Cohort
All-Cause Mortality (participants affected / at risk) | 14/274 | 8/63 | 2/45
Serious Adverse Events (participants affected / at risk) | 175/274 | 42/63 | 24/45
Other Adverse Events (participants affected / at risk) | 176/274 | 34/63 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Cohort (N=274) | Roll-In Cohort (N=63) | Bicuspid Cohort (N=45)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0 | 0
Accelerated idioventricular rhythm (Cardiac disorders) | 1 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 3 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 5 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 12 | 5 | 2
Atrial flutter (Cardiac disorders) | 2 | 1 | 0
Atrioventricular block (Cardiac disorders) | 4 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 61 | 17 | 6
Atrioventricular block first degree (Cardiac disorders) | 3 | 2 | 1
Atrioventricular block second degree (Cardiac disorders) | 7 | 0 | 2
Bradycardia (Cardiac disorders) | 3 | 0 | 0
Bundle branch block left (Cardiac disorders) | 36 | 7 | 7
Cardiac arrest (Cardiac disorders) | 4 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 3 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 15 | 5 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Chordae tendinae rupture (Cardiac disorders) | 1 | 0 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 4 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 2 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0
Paravalvular aortic regurgitation (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 7 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 3 | 1 | 1
Sinus arrest (Cardiac disorders) | 2 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 2 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 1 | 0
Blindness (Eye disorders) | 1 | 0 | 0
Open angle glaucoma (Eye disorders) | 1 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0
Retinal infarction (Eye disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Cardiac complication associated with device (General disorders) | 0 | 0 | 1
Catheter site haematoma (General disorders) | 3 | 0 | 0
Catheter site haemorrhage (General disorders) | 2 | 0 | 1
Death (General disorders) | 3 | 0 | 1
Device embolisation (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 2 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Structural valve deterioration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 1 | 0
Echocardiogram abnormal (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 2 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Alcoholic seizure (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 3 | 1
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 7 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 1 | 0
Mononeuropathy (Nervous system disorders) | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 3 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 5 | 0 | 0
Device failure (Product Issues) | 2 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 3 | 2
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Ovarian mass (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 5 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 2 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 2 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Cohort (N=274) | Roll-In Cohort (N=63) | Bicuspid Cohort (N=45)
Leukocytosis (Blood and lymphatic system disorders) | 6 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 3 | 5
Atrial fibrillation (Cardiac disorders) | 25 | 4 | 6
Atrioventricular block first degree (Cardiac disorders) | 18 | 0 | 2
Bundle branch block left (Cardiac disorders) | 90 | 18 | 13
Nausea (Gastrointestinal disorders) | 2 | 0 | 3
Non-cardiac chest pain (General disorders) | 5 | 2 | 3
Headache (Nervous system disorders) | 1 | 0 | 3
Hypotension (Vascular disorders) | 12 | 5 | 3

LIMITATIONS AND CAVEATS:
The study was terminated during enrollment and all follow-up of patients was also discontinued. As a result, the primary outcome is not representative of the full cohort of patients and represents a significantly smaller sample of patients to reach the 1 year timepoint in the Main cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PI and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/95/NCT03618095/Prot_SAP_000.pdf